CLINICAL TRIAL: NCT05467098
Title: Does Dry Needling Change Shoulder Muscle Blood Flow, Motions, and Pain Sensitivity?
Brief Title: Dry Needling and Shoulder Muscle Blood Flow, Motions, and Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Jace Brown, Principal Investigator, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY2022-349
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dry Needling; Shoulder Pain
Keywords: shoulder pain; dry needling; pain pressure threshold
MeSH Terms: conditions — Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Pre-test post-test Design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individuals with and without Shoulder Pain (Experimental): Individuals with shoulder pain will receive dry needling to the two to four most tender points in the infraspinatus based on examiner palpation
  Individuals without shoulder pain will receive dry needling to two points in the muscle belly of the infraspinatus near the insertion and below the midpoint of the spine of the scapula
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the MTrP of the infraspinatus muscles. Once the needle has been inserted, the technique described by Hong (1994) will be used. The needle will be pistoned in an up and down motion within the infraspinatus muscle at approximately 1Hz for 10 seconds with the aim of eliciting local twitch responses.

SUMMARY:
Shoulder pain is one of the most common reasons people consult with their primary health care provider, and 40-50% of these patients with shoulder pain continued to complain of persistent symptoms after 6 to 12 months. It has been suggested that the presence of myofascial trigger points (MTrPs) may contribute to the chronicity of shoulder symptoms. An MTrP is a hyperirritable taut band of tissue within a muscle that produces pain when stimulated MTrPs are common in patients with shoulder disorders and occur most often in the infraspinatus muscle of a painful shoulder MTrPs were associated with an acidic biochemical environment with elevated levels of inflammatory mediators, neuropeptides, and proinflammatory cytokines such as bradykinin and calcitonin g-related peptide. It was hypothesized that metabolic demands on muscle and capillary constrictions may contribute to the development of MTrPs. To date, only a few studies have examined the vascular environment of MTrPs and surrounding areas before and after dry needling. No studies have yet examined whether dry needling would change blood flow in patients with shoulder pathology. Therefore, the purpose of this pilot study is to examine the effect of dry needling on blood flow of the infraspinatus muscle using color Doppler imaging in individuals with and without shoulder pain.

DETAILED DESCRIPTION:
RESEARCH DESIGN

The research design for this experimental study will be a repeated measures design. The outcome variables collected in this study are the following: peak systolic velocity, end diastolic velocity, resistive index, pulsatile index, of the infraspinatus, shoulder range of motion (ROM) of internal and external rotations, and Pain pressure threshold (PPT).

PROCEDURE

Eligible participants will be asked to complete an intake form (see Section 6 and 9), asking them about their demographic data, including age, gender, height, weight, occupation, past medical history, and questions related to their shoulder pain (onset, injury mechanism if any, location, duration, type, and nature). The participant's eligibility will be confirmed by the Principal Investigator (PI). Next, each participant will complete the shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH) to determine the participants disability level due to their shoulder pain. After gathering the subjective information and confirming presence of MTrP using palpation, blood flow parameters, shoulder ROMs and PPTs will be collected from the most painful side. If both sides are equally painful, a coin-flip will be used to determine the side of testing. In a subgroup of the first 15 participants in each group, the outcome measures will be assessed twice with a 5-minute break between each measure to establish the reliability prior to the dry needling intervention. The outcome measurements will be administered in an order of shoulder ROMs, followed by PPT and blood flow parameters before the dry needling and in a reverse order of blood flow parameters, PPT and shoulder ROM after dry needling in order to minimize the position changes and to capture immediate changes of blood flow.

SHOULDER RANGE OF MOTION

Range of motion testing will be performed with the individual in supine with the shoulder at 90° abduction and 10° of horizontal abduction with 90° of elbow flexion. Two examiners (The PI and a research assistant) will be responsible for all the measurements, one to measure the shoulder ROM and the other to read the measurements off the goniometer. The center of rotation of the goniometer will be placed over the olecranon while one arm of the goniometer will be positioned along the length of the ulna, aligned with the ulnar styloid process. The other arm will be positioned perpendicular to the ground. For both measurement of shoulder internal and external rotation, scapular compensation will be monitored by using the thumb on the coracoid process and fingers along the spine of the scapula. Each measurement will be repeated three times with the average measurements used for data analysis.

PRESSURE PAIN THRESHOLD TESTING

During the PPT testing, the participant will be placed in the prone position with upper extremities relaxed at their sides. PPT of the infraspinatus will be tested in the muscle belly below the midpoint of the spine of scapula. The participants will be given a stop button and instructed to stop the test as soon as the pressure becomes uncomfortable or painful, and not to allow a painful or uncomfortable sensation to continue. The participants will be familiarized with the algometer, which will consist of a single trial on the non-painful side to ensure that the participant understands the process. An average of three trials will be used for data analysis.

ULTRASOUND IMAGING

Each participants will remain in the same position for ultrasound imaging. The ultrasound transducer will be placed perpendicular to the infraspinous fossa to visualize arterioles or arteries in the vicinity of the MTrPs and to quantify the velocity of blood flow at the MTrPs of the infraspinatus determined by palpation by the PI (JB) during the eligibility screen. The location of the transducer will be outlined after initial placement to ensure consistent placement of the transducer between the testing sessions. The spectral Doppler waveforms will be analyzed to trace the velocities throughout the cardiac cycle. The peak systolic (PSV), end diastolic velocity (EDV), resistive index (RI) and pulsatile index (PI) will be calculated using software available on the device. On a Doppler waveform, the PSV corresponds to each "peak" within the spectral window, whereas the EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak. These values will be used to calculate the RI with the formula RI = (PSV - EDV)/PSV and the PI with the formula PI = (PSV - EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle.

INTERVENTION

Following the baseline testing, the PI will perform the dry needling intervention. A sterile, disposable, solid filament needle (Seirin Corp., Shizuoka, Japan) will be inserted manually into the MTrP of the infraspinatus muscle. Once the needle has been inserted, the needle will be pistoned in an up-and-down motion within the infraspinatus muscle at approximately 1Hz for 10 seconds, Individuals with shoulder pain will receive dry needling to the two to four most tender points in the infraspinatus based on examiner palpation (JB). The control group will receive dry needling to two points in the muscle belly of the infraspinatus near the insertion and below the midpoint of the spine of the scapula.

REASSESSMENT

Immediately following the interventions, measures of the three outcomes will be collected in the following order to minimize position changes for all participants (blood flow parameters, infraspinatus PPT, and shoulder range of motion). Additionally, any adverse events following the dry needling procedures will be assessed immediately, such as bruising, nausea, dizziness, or post-needling soreness. If bleeding occurs, the participant will be informed.

ELIGIBILITY:
Inclusion Criteria:

Individuals without shoulder pain:

* Ages 18-65 and without a history of shoulder pain in the last 12 months
* absence of a MTrP in the infraspinatus as determined by palpation

Individuals with shoulder pain:

* Ages 18-65 with unilateral nonspecific shoulder pain based on participants' self-reported pain level of greater than or equal to 2/10 on the Numeric Pain Rating Scale (NPRS) in last 24 hours
* non-traumatic origin of pain
* presence of at least one MTrP with referral pain pattern in the infraspinatus muscle determined through palpation.

Exclusion Criteria:

* systemic joint disease (e.g. rheumatoid arthritis)
* evidence of red flags (e.g. fracture, infection, tumor, cauda equina syndrome)
* cancer
* neurological disorders
* neuropathy
* Raynaud's disease
* pregnancy
* previous shoulder surgery
* repeated infection
* immunocompromised disease (e.g., diabetes mellitus, HIV, AIDS, lupus)
* inability to maintain the testing and treatment positions (i.e., supine and prone-lying) for 15 minutes at a time.
* bleeding disorders (e.g. hemophilia)
* use of anti-coagulants (e.g. Coumadin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity (PSV) | Change from baseline PSV immediately
  On a Doppler waveform, the PSV corresponds to each "peak" within the spectral window. These values will be used to calculate the RI with the formula RI = (PSV - EDV)/PSV.
End Diastolic Velocity (EDV) | Change from baseline EDV immediately
  EDV corresponds to the point marked at the end of the cardiac cycle just prior to the systolic peak.
Resistive Index (RI) | Change from baseline RI immediately
  Resistive Index is used to assess the resistance in a pulsatile vascular system.The RI is defined by the the formula RI = (PSV - EDV)/PSV.
Pulsatile Index (PI) | Change from baseline PI immediately
  Pulsatility index (PI) is defined as the difference between the peak systolic flow and minimum diastolic flow velocity, divided by the mean velocity recorded throughout the cardiac cycle. It is a non-invasive method of assessing vascular resistance with the use of Doppler ultrasonography. PI is defined with the formula PI = (PSV - EDV)/mean velocity, where mean velocity is the average flow velocity during the cardiac cycle.

SECONDARY OUTCOMES:
Pain Pressure Thresholds | Change from baseline Pain Pressure Threshold immediately
  Pressure pain threshold (kPa) is a quantitative sensory test, used to measure deep muscular tissue sensitivity to mechanical pressure stimuli. The test determines the amount of pressure over the infraspinatus in which a steadily increasing non-painful pressure stimulus turns into a painful pressure sensation.
Shoulder Range of Motion | Change from baseline shoulder range of motion immediately
  shoulder range of motion of internal and external rotation is the number of degrees of motion measured using standard goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jace A Brown, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the summary data are published. Data obtained through this study may be provided to qualified researchers with academic interest in Dry Needling. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Bron C, Dommerholt J, Stegenga B, Wensing M, Oostendorp RA. High prevalence of shoulder girdle muscles with myofascial trigger points in patients with shoulder pain. BMC Musculoskelet Disord. 2011 Jun 28;12:139. doi: 10.1186/1471-2474-12-139. PMID 21711512
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Diaz-Rodriguez L, Gonzalez-Iglesias J, Palacios-Cena D, Arroyo-Morales M. Changes in pain and pressure pain sensitivity after manual treatment of active trigger points in patients with unilateral shoulder impingement: a case series. J Bodyw Mov Ther. 2011 Oct;15(4):399-404. doi: 10.1016/j.jbmt.2010.12.003. Epub 2011 Jan 17. PMID 21943613
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] de Micco C, Toga M. [The immune status of the central nervous system]. Rev Neurol (Paris). 1988;144(12):776-88. French. PMID 3070691
- [Background] Sandberg M, Lundeberg T, Lindberg LG, Gerdle B. Effects of acupuncture on skin and muscle blood flow in healthy subjects. Eur J Appl Physiol. 2003 Sep;90(1-2):114-9. doi: 10.1007/s00421-003-0825-3. Epub 2003 Jun 24. PMID 12827364
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Nascimento JDSD, Alburquerque-Sendin F, Vigolvino LP, Oliveira WF, Sousa CO. Absolute and Relative Reliability of Pressure Pain Threshold Assessments in the Shoulder Muscles of Participants With and Without Unilateral Subacromial Impingement Syndrome. J Manipulative Physiol Ther. 2020 Jan;43(1):57-67. doi: 10.1016/j.jmpt.2019.04.002. Epub 2020 Feb 13. PMID 32061418